CLINICAL TRIAL: NCT05014386
Title: Ahmed Glaucoma Valve Implantation With Ologen Augmentation in Secondary Pediatric Glaucomas
Brief Title: AGV Implantation With Ologen in Pediatric Glaucomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Associate professor of ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGV with ologen in SPG
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma
Keywords: Ahmed Glaucoma Valve; Ologen; secondary pediatric glaucomas
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, controlled couple armed study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ahmed Glaucoma Valve Implantation (Active Comparator): A 7-0 silk traction suture was placed through the clear cornea.A conjunctival incision was made 4 mm posterior to the limbus in the supratemporal quadrant. After dissecting conjunctiva and Tenon's primed FP7 or FP8 AGV was inserted into the subconjunctival space and sutured to sclera using two interrupted 7-0 silk sutures 8-10 mm posterior to the limbus. A 23-gauge needle was used to enter the anterior chamber from the surgical limbus. The tube then was cut beveled up and inserted into the anterior chamber through the tunnel. Finally, conjunctiva and Tenon were approximated using a running 8-0 Vicryl suture.At the close of surgery, subtenon antibiotic and steroids were injected in all cases.
  Interventions: Procedure: Ahmed Glaucoma Valve Implantation in secondary pediatric glaucomas.
- Ologen augmentation group (Active Comparator): In addition to what is planned for the other Arm;, a round 12 × 1 mm circular Ologen disc will be placed over the FP7 or FP8 AGV-plate immediately before conjunctival closure.
  Interventions: Procedure: Ahmed Glaucoma Valve Implantation with Ologen augmentation in secondary pediatric glaucomas

INTERVENTIONS:
Procedure: Ahmed Glaucoma Valve Implantation in secondary pediatric glaucomas. — A 7-0 silk traction suture was placed through the clear cornea.A conjunctival incision was made 4 mm posterior to the limbus in the supratemporal quadrant. After dissecting conjunctiva and Tenon's primed FP7 or FP8 AGV was inserted into the subconjunctival space and sutured to sclera using two interrupted 7-0 silk sutures 8-10 mm posterior to the limbus. A 23-gauge needle was used to enter the anterior chamber from the surgical limbus. The tube then was cut beveled up and inserted into the anterior chamber through the tunnel. Finally, conjunctiva and Tenon were approximated using a running 8-0 Vicryl suture.At the close of surgery, subtenon antibiotic and steroids were injected in all cases.
  Arms: Ahmed Glaucoma Valve Implantation
Procedure: Ahmed Glaucoma Valve Implantation with Ologen augmentation in secondary pediatric glaucomas — A 7-0 silk traction suture was placed through the clear cornea.A conjunctival incision was made 4 mm posterior to the limbus in the supratemporal quadrant. After dissecting conjunctiva and Tenon's primed FP7 or FP8 AGV was inserted into the subconjunctival space and sutured to sclera using two interrupted 7-0 silk sutures 8-10 mm posterior to the limbus. A 23-gauge needle was used to enter the anterior chamber from the surgical limbus. The tube then was cut beveled up and inserted into the anterior chamber through the tunnel. a round 12 × 1 mm circular Ologen disc will be placed over the FP7 or FP8 AGV-plate immediately before conjunctival closure. Finally, conjunctiva and Tenon were approximated using a running 8-0 Vicryl suture.At the close of surgery, subtenon antibiotic and steroids were injected in all cases.
  Arms: Ologen augmentation group

SUMMARY:
Ahmed Glaucoma Valve Implantation with Ologen augmentation in secondary pediatric glaucomas: A 2-year randomized controlled trial.

Background:

Many studies have investigated the clinical benefits of Ologen for trabeculectomy. However, its benefits for Ahmed glaucoma valve implantation have not been widely investigated.

Purpose:

The aim of this study was to compare the 2-year outcomes of AGV implantation with and without Ologen adjuvant for the treatment of children with 2ry pediatric glaucoma. Design: This is a single-center, randomized, controlled study. Participants: Consecutive children with refractory pediatric glaucoma requiring AGV implantation were enrolled in this study.

Methods:

Refractory pediatric glaucoma was defined by at least 2 repeated IOP measurements greater than 21 mmHg and accompanying signs of buphthalmos, corneal edema, Haabs striae, or optic nerve cupping despite maximal tolerated medical therapy. The primary outcome measure was AGV success. Complete success was defined as intraocular pressure (IOP) between 6 and 20 mmHg without glaucoma medications and additional IOP-lowering surgeries. Qualified success was defined as above, except IOP control maintained with glaucoma medications. In Ologen eyes, a round 12 × 1 mm circular Ologen disc will be placed over the FP7 or FP8 AGV-plate immediately before conjunctival closure. Control eyes received conventional FP7 or FP8 AGV surgery without Ologen augmentation.

DETAILED DESCRIPTION:
Ahmed Glaucoma Valve Implantation with Ologen augmentation in secondary pediatric glaucomas: A 2-year randomized controlled trial.

Background:

The management of secondary pediatric glaucoma is challenging in terms of maintaining lifelong vision and avoiding an aggressive scarring course after surgery. Secondary Pediatric glaucoma includes a variety of ocular conditions that lead to high intraocular pressure (IOP) and progressive optic neuropathy. Glaucoma is a well-known complication of congenital cataract extraction and is the most frequent long-term complication of lensectomy with or without intraocular lens (IOL) implantation. The reported incidence in the literature is between 15% and 45%4. Another cause is aphakic glaucoma.Management of secondary pediatric glaucoma is mainly surgical, and medical therapy is used either as a temporizing measure or as an adjunctive treatment.

Traditionally, "staged approach" has been favored by many ophthalmologists. This involves starting with angle surgeries and their repetition in the case of failure, proceeding with trabeculectomy or combined trabeculotomy-trabeculectomy for refractory patients, and drainage device or cyclodestruction for very advanced patients.The poor clinical outcomes prompted surgeons to adapt glaucoma drainage devices (GDDs) as a mainstay of treatment for refractory glaucoma in both pediatric and adult populations.In children, Ahmed glaucoma valves (AGV) have greater than 80% success rate at 1- year, but success decreases to less than 50% by 5 years2. In order to improve long-term IOP control, mitomycinC (MMC) has been used as an adjuvant during implant placement. While MMC is a commonplace in trabeculectomy, its use with GDDs is controversial due to increased complications such as bleb leaks and endothelial cell damage. More recently, Ologen, a biodegradable Type-I collagen matrix, has been used in glaucoma surgeries. Ologen is safe and effective in enhancing trabeculectomy surgery in adults and children,.

Many studies have investigated the clinical benefits of Ologen for trabeculectomy. However, its benefits for Ahmed glaucoma valve implantation have not been widely investigated. Reports in adult patients have shown that Ologen may increase AGV success and decrease hypertensive phase incidence. Many studies have investigated the clinical benefits of Ologen for trabeculectomy. However, its benefits for Ahmed glaucoma valve implantation have not been widely investigated. As glaucoma drainage devices are being increasingly used for pediatric glaucoma,investigators decided to report the results and safety of Ahmed glaucoma valve (AGV) implantation in a series of secondary pediatric glaucoma as well as the clinical benefits of concomitant use Ologen as an adjuvant for for Ahmed glaucoma valve implantation .

Purpose:

The aim of this study was to compare the 2-year outcomes of AGV implantation with and without Ologen adjuvant for the treatment of children with 2ry pediatric glaucoma.

Design:

This is a single-center, randomized, controlled study.

Participants:

Consecutive children with refractory pediatric glaucoma requiring AGV implantation were enrolled in this study.

Methods:

Refractory pediatric glaucoma was defined by at least 2 repeated IOP measurements greater than 21 mmHg and accompanying signs of buphthalmos, corneal edema, Haabs striae, or optic nerve cupping despite maximal tolerated medical therapy. The primary outcome measure was AGV success. Complete success was defined as intraocular pressure (IOP) between 6 and 20 mmHg without glaucoma medications and additional IOP-lowering surgeries. Qualified success was defined as above, except that IOP control was maintained with glaucoma medications.

Surgical procedure:

A 7-0 silk traction suture was placed through the clear cornea.A conjunctival incision was made 4 mm posterior to the limbus in the supratemporal quadrant. After dissecting conjunctiva and Tenon's primed FP7 or FP8 AGV was inserted into the subconjunctival space and sutured to sclera using two interrupted 7-0 silk sutures 8-10 mm posterior to the limbus. A 23-gauge needle was used to enter the anterior chamber from the surgical limbus. The tube then was cut beveled up and inserted into the anterior chamber through the tunnel. In Ologen eyes, a round 12 × 1 mm circular Ologen disc will be placed over the FP7 or FP8 AGV-plate immediately before conjunctival closure. Control eyes received conventional FP7 or FP8 AGV surgery without Ologen augmentation.

Finally, conjunctiva and Tenon were approximated using a running 8-0 Vicryl suture.At the close of surgery, subtenon antibiotic and steroids were injected in all cases.

Data collection:

Preoperative data including age at the time of surgery, sex,laterality, type of glaucoma, prior ocular history, prior surgical treatment, number of glaucoma medications, IOP, cup to disc ratio, and central corneal thickness (CCT) were extracted from patients' record. Postoperative data included follow-up durations; IOP at months 3, 6, 12, 24, and 36; cup to disc ratios at months 12, 24,; and intraoperative and postoperative complications. In all cases, IOPs were measured by Tono-Pen (Mentor, Woburn, MA, USA) under anesthesia. In the clinic, IOPs were measured by ICare (ICare Finland Oy, Helsinki, Finland) and Goldmann applanation tonometer (Haag-Streit, Köniz, Switzerland).

Statistical analysis:

All statistical analysis was accomplished using IBM SPSS version 20. Assessment of the data normality was done using both Histogram plot and Shapiro-Wilk's test. Wilcoxon test was used to compare the preoperative and postoperative variables in each group. The comparison between the two groups was done using Mann-Whitney test for numerical variables and Chi-square test for categorical variables. Kaplan-Meier survival curve was plotted to estimate the mean survival time and probabilities of failure at different follow-up stages in the both groups. For all tests, P value of less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Refractory pediatric glaucoma was defined by at least 2 repeated IOP measurements greater than 21 mmHg and accompanying signs of buphthalmos, corneal edema, Haabs striae, or optic nerve cupping despite maximal tolerated medical therapy.

Exclusion Criteria:

* Primary congenital glaucoma

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
AGV success | 2 years
  Complete success was defined as intraocular pressure (IOP) between 6 and 20 mmHg without glaucoma medications and additional IOP-lowering surgeries. Qualified success was defined as above, except that IOP control was maintained with glaucoma medications.

SECONDARY OUTCOMES:
cup to disc ratios | 2 years
  cup to disc ratio
postoperative complications | 2 years
  postoperative complications

IPD SHARING:
Plan to Share IPD: Yes
The (IPD) will be provided as supplemental digital content
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: IPD will be provided with publications as supplementary digital content